CLINICAL TRIAL: NCT05958654
Title: Detection of Elder Mistreatment Through Emergency Care Technicians - Revised for Primary Care (DETECT-RPC) Universal EM Screening
Brief Title: DETECT-RPC Universal EM Screening
Acronym: DETECT-RPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Bradley Cannell, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: DETECT-RPC; 4R33AG078523-03 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Elder Abuse; Elder Mistreatment
Keywords: Elder Mistreatment
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with DETECT-RPC screening tool (Experimental)
  Interventions: Behavioral: Detection of Elder mistreatment Through Emergency Care Technicians-Revised for Primary Care (DETECT-RPC) screening tool
- without DETECT-RPC screening tool (No Intervention)

INTERVENTIONS:
Behavioral: Detection of Elder mistreatment Through Emergency Care Technicians-Revised for Primary Care (DETECT-RPC) screening tool — DETECT is an elder mistreatment (EM) screening tool created for medics in the Fort Worth Texas area to use when responding to the homes of older adults, enabling them to screen for signs of elder mistreatment. DETECT-RPC is the adapted version of this tool designed specifically for use by home-based primary care (HBPC) clinicians.
  The DETECT-RPC tool is designed to:
  1. Be brief and easy to use.
  2. Focus on the clinician's direct observations of the older adult and their physical and social environment.
  3. Provide clear guidance on reporting suspected EM.
  4. Integrate seamlessly into existing procedures and medical charting systems.
  Other Names: DETECT-RPC screening tool
  Arms: with DETECT-RPC screening tool

SUMMARY:
The purpose of this study is to evaluate whether the use of the Detection of Elder Mistreatment Through Emergency Care Technicians-Revised for Primary Care (DETECT-RPC) screening tool increases the average reporting of elder mistreatment (EM) by homebased primary care (HBPC) clinicians.

ELIGIBILITY:
Inclusion Criteria (Clinicians):

* Clinician who actively provides home-based primary care (HBPC) to patients enrolled in one of our partner home-based primary care programs at least part time.

Exclusion Criteria (Clinicians):

* HBPC Clinicians must be a physician, nurse practitioner, or physician assistant who actively provides home-based primary care to patients enrolled at a partner site HBPC at least part time

Inclusion Criteria (patients):

* in home-based primary care
* 60 years or older
* seen by a clinician participating in the study

Exclusion Criteria (patients)

* Must be aged 60 and older, enrolled in a site-specific partner HBPC and treated in their primary residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
number of reports of EM | from randomization to termination of data collection (3 years)
  Data will be collected on the number of reports of EM made by clinicians to the appropriate authorities [for example, adult protective services (APS)]
Mortality | from randomization to termination of data collection (3 years)
  Mortality among patients will be assessed among patients enrolled in the partner home-based primary care programs.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Cannell, PhD,MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - John Hopkins University Medicine International, Baltimore, Maryland
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas health Science Center at Houston( LBJ House Calls Program), Houston, Texas
  - The University of Texas Health Science Center at Houston( UT Physicians House Calls Program), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cannell B, Sevey N, Livingston MD, Burnett J, Lees Haggerty K, Pickering C. Detection of Elder Abuse Through Emergency Care Technicians Screening Tool Revision for Home-Based Primary Care (DETECT-RPC): a cluster randomised controlled trial study protocol. BMJ Open. 2025 Jan 15;15(1):e089028. doi: 10.1136/bmjopen-2024-089028. PMID 39819945